CLINICAL TRIAL: NCT00783250
Title: Effect of Bronchodilators on Respiratory Mechanics in COPD Patients With Poor Reversibility
Brief Title: Bronchodilators and Respiratory Mechanics in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Problems with data collection
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Chief ICU, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 350
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Respiratory Mechanics; Bronchodilators; COPD patients with poor reversibility
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salbutamol+Tiotropium (Experimental): Salbutamol will be given at the dose of 400 micrograms and Tiotropium at the dose of 18 micrograms
  Interventions: Drug: Salbutamol + Tiotropium
- placebo + Tiotropium (Placebo Comparator): Placebo using MDI + administration of Tiotropium after 20 minutes
  Interventions: Drug: Placebo + Tiotropium

INTERVENTIONS:
Drug: Salbutamol + Tiotropium — Salbutamol 400 micrograms + Tiotropium 18 micrograms
  Other Names: Ventolin; Spiriva
  Arms: Salbutamol+Tiotropium
Drug: Placebo + Tiotropium — Placebo via MDI + Tiotropium 18 micrograms
  Other Names: Spiriva
  Arms: placebo + Tiotropium

SUMMARY:
The aim of this study is to assess the effects on respiratory mechanics of one "classical" short-term bronchodilator (i.e., salbutamol) versus placebo, and to verify the hypothesis that the addition of another bronchodilator (i.e., anticholinergic) may induce a further improvement on the work of breathing of stable COPD patients.

DETAILED DESCRIPTION:
Studies with long-acting b2-agonists in COPD patients who poorly respond to routine airways obstruction reversibility tests with forced expiratory manoeuvres, such as forced expiratory volume in one second (FEV1), are scarce. Such studies, however, seem to show favourable effects on clinical parameters.

This may explain the subjective improvements and changes in quality of life with long-acting b2-agonists in patients with COPD. The lack of effect on forced expiration tests may be due to early airway collapse and subsequent airflow decline causing underestimation of the existing bronchodilatory effects located more peripherally in the respiratory tract, where the major site of resistance is located in obstructive lung disease.

We therefore design a study aimed to assess the short term effects of one short-acting beta2-agonist vs placebo, and the effects of an additional and sequential administration of a different bronchodilator, like tiotropium bromide (anticholinergic agent) on the work of breathing, and its components (i.e., lung resistances and compliance) of COPD patients with poor reversibility assessed using the classical Pulmonary Function Tests.

ELIGIBILITY:
Inclusion Criteria:

* COPD patient with a Tiffenau ratio <55% and >25% predicted
* Poor reversibility to an acute bronchodilator test (i.e. FEV1 changes<10% from baseline)

Exclusion Criteria:

* Lack of informed consent
* Cancer
* Concomitant lung and airways diseases

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Recordings of respiratory mechanics | 90 minutes

SECONDARY OUTCOMES:
Dyspnea score | 90 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Unit Fondazione S.Maugeri, Pavia, PV, Italy